CLINICAL TRIAL: NCT02246595
Title: A Phase II Randomized, Placebo-controlled, Double-blind, Dose Controlled Trial in Patients Suffering From Early, Newly Developing Abdominal or Pulmonary Derived Septic Organ Dysfunction to Evaluate Safety, Pharmacokinetics, Pharmacodynamics and to Estimate Efficacy of the New Humanized Monoclonal i.v. Administered Antibody CaCP29
Brief Title: Studying Complement Inhibition in Early, Newly Developing Septic Organ Dysfunction
Acronym: SCIENS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InflaRx GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IFX-1-P2.1; 2013-001037-40 (EudraCT Number)
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Sepsis; Severe Sepsis; Septic Shock; Systemic Inflammatory Response Syndrome; Organ Dysfunction
MeSH Terms: conditions — Sepsis; Shock, Septic; Systemic Inflammatory Response Syndrome | interventions — vilobelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CaCP29 (Active Comparator): dose escalating i.v. administration of CaCP29 (verum)
  Interventions: Biological: CaCP29
- Placebo (Placebo Comparator): dose escalation mimicing i.v. placebo treatment:
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CaCP29
  Other Names: IFX-1
  Arms: CaCP29
Biological: Placebo
  Arms: Placebo

SUMMARY:
The trial enrolls patients with early severe sepsis or septic shock displaying at least one newly developed organ dysfunction and showing clinical evidence of pulmonary or abdominal infection. The primary goal of the trial is to assess the pharmacokinetics and pharmacodynamics of the new monoclonal antibody CaCP29 and to characterize safety and tolerability as well as evaluate parameters of efficacy.

ELIGIBILITY:
Key Inclusion Criteria at screening:

1. Male or female patients >= 18 years old
2. Written informed consent
3. Occurrence of at least two criteria of a systemic inflammatory response syndrome (SIRS) not explained by other reasons. These criteria should be present within 12 hours prior to screening
4. Suspected or confirmed abdominal or pulmonary infection at screening
5. Broad spectrum i.v. antimicrobial therapy to treat abdominal or pulmonary infection
6. At least one of the following acute organ dysfunctions due to sepsis. Each organ dysfunction must have occurred within 12 hours prior to screening, cannot mainly be explained by other disease processes than sepsis and is judged by the investigator as being caused or directly related to an abdominal or pulmonary infectious focus:

   1. respiratory
   2. renal
   3. hematologic
   4. metabolic
   5. cardiovascular (occurred within the last three hours)
7. Reasonable likelihood that administration of study drug can be started within 3.5 hours after start of screening process

Key Exclusion Criteria at screening:

1. Sepsis of other primary cause than pulmonary or abdominal source
2. Weight > 130 kg at screening
3. Any other disease and condition that is likely to interfere with evaluation of study product, outcome assessment or satisfactory conduct of the study
4. Patients receiving the following concomitant medication within 14 days prior to screening:

   1. Calcineurin inhibitors (e.g., ciclosporine, tacrolimus)
   2. Proliferation inhibitors (e.g., everolimus, sirolimus)
   3. Anti-metabolites (e.g., mycophenolate, mycophenolic acid, azathioprine)
   4. High dose corticosteroids (e.g., > 50mg prednisolon per day or equivalent)
5. Patients receiving high dose immunoglobulins within 3 months prior to screening
6. Patients with following abnormal laboratory result: Neutrocytopenia with neutrophil count < 1,000/mm3 unless likely due to sepsis
7. General criteria:

   1. Pregnant (in women of childbearing potential an urine pregnancy test has to be performed) or breast-feeding women
   2. Women with childbearing potential (defined as within two years of their last menstruation) not willing to practice appropriate contraceptive measures (e.g., implanon, injections, oral contraceptives, intrauterine devices, partner with vasectomy, abstinence) while participating in the trial
   3. Participation in any interventional clinical trial within the last three months
   4. Prior participation in this clinical trial
   5. Patient is chronically bed-bound prior to the onset of sepsis
   6. Known intravenous drug abuse
   7. Employee at the study site, spouse/partner or relative of any study staff (e.g., investigator, sub-investigators, or study nurse) or relationship to the sponsor
   8. No commitment to full aggressive life support (e.g., do not resuscitate order)

Inclusion Criteria at randomisation:

1. At least one of the sepsis related organ dysfunction detected at screening is still present
2. Current treatment with broad spectrum i.v. antibiotics has been started or is ongoing

Exclusion Criteria at randomisation:

1. Time frame between detection of a non cardiovascular organ dysfunction and start of randomization procedure is more than 15 hours
2. Time frame between detection of a cardiovascular organ dysfunction and start of randomization is more than six hours
3. Organ dysfunctions are unlikely to be persistent for next three hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of CaCP29 | 0h, 2h, 6h, 12h, 14h (only cohort 1), 24h, 26h (only cohort 2 and 3), 48h, 72h, 74h (only cohort 3), days 5, 8, 13, 28
  Pharmacokinetic measures include
  * Plasma concentration over time
  * Maximum observed concentration per infusion
  * Concentration measured immediately before next dosing
  * Area under the curve of plasma concentration per infusion
  * Mean concentration per infusion
  * Terminal phase half-life
Assess the pharmacodynamic (PD) effects of CaCP29 on the change from baseline in plasma concentrations of C5a | 0h, 2h, 6h, 12h, 14h (only cohort 1), 24h, 26h (only cohort 2 and 3), 48h, 72h, 74h (only cohort 3), days 5, 8, 13, 28
Safety variables will be summarized using descriptive statistics based on adverse event collection | 28 days

SECONDARY OUTCOMES:
Anti-drug antibodies (ADA) | 28 days or hospital discharge
  The development of ADA will be described by:
  * Number of patients with detection of anti-drug antibody (ADA)
  * Number of patients with detection of ADA at each time point measured
All-cause mortality rate | 28 days
Morbidity | daily
  * Mean SOFA until Day 10
  * Modified mean SOFA until day 10 (calculated by omitting the Central Nervous System sub-score and calculating the renal subscore without taking urine output into consideration)
  * Mean SOFA Sub-scores until Day 10
  * Days on ICU until Day 28
  * Number of patients ventilated until Day 14
  * Ventilator-free days until Day 14
  * Numbers of patients with renal replacement therapy (RRT) until Day 14
  * RRT-free days until Day 14
  * Numbers of patients with administration of vasopressor until Day 14
  * Vasopressor-free days until Day 14
  * Days without antimicrobial therapy (AMT) until Day 14
Fluid balance | 28 days or ICU discharge
  * Mean daily total fluid intake until Day 28 (maximal until ICU discharge)
  * Mean daily total fluid output until Day 28 (maximal until ICU discharge)
  * Mean daily fluid balance until Day 28 (maximal until ICU discharge)
Change in routine laboratory parameters as compared to baseline | Days 1, 2, 3, 4, 5, 8, 13, 28
Change in ECG as compared to baseline | Days 2, 4, 8, 28
Change in vital signs as compared to baseline | Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bauer, Prof. Dr., Principal Investigator — University Hospital Jena
Locations (11):
- Germany (11):
  - Study Site, Aachen
  - Study Site, Augsburg
  - Study Site, Bad Saarow
  - Study Site, Berlin
  - Study Site, Göttingen
  - Study Site, Greifswald
  - Study Site, Hamburg
  - Study Site, Jena
  - Study Site, Kiel
  - Study Site, Leipzig
  - Study Site, Oldenburg